CLINICAL TRIAL: NCT04441398
Title: Prospective, Randomized, Double-blind, Parallel, Placebo Controlled Study to Evaluate the Safety and Efficacy of Nitazoxanide 600 mg to Treat Ambulatory Adult Subjects Diagnosed With COVID-19 With Mild Symptoms Assisted in the Public Health System of the City of Mesquita
Brief Title: Efficacy and Safety of Nitazoxanide 600 mg to Treat Mild Ambulatory COVID-19 Patients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's strategic decision
Sponsor: Azidus Brasil (Industry)
Collaborators: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NITFQM0720OR
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: covid19
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either nitazoxanide (n=150) or placebo (n=150)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nitazoxanide (Experimental): Subjects will receive nitazonanide 600 mg TID.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Subjects will receive placebo TID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Subjects will receive nitazonanide 600 mg TID for 7 days. Treatment can be extended for another 7 days at Investigators discretion.
  Other Names: Viranitta
  Arms: nitazoxanide
Drug: Placebo — Subjects will receive placebo TID for 7 days. Treatment can be extended for another 7 days at Investigators discretion.
  Arms: Placebo

SUMMARY:
The aim is to demonstrate a decrease in complications among ambulatory patients who are diagnosed with mild COVID-19 by treating them with nitazoxanide for 7 to 14 days on top of standard care compared to patients who receive standard care and placebo only.

DETAILED DESCRIPTION:
The aim is to demonstrate a decrease in complications among ambulatory patients who are diagnosed with mild COVID-19 by treating them with nitazoxanide for 7 to 14 days on top of standard care compared to patients who receive standard care and placebo only.

After 7 days of treatment, the Investigator can extend the treatment duration for another 7 days at his/her discretion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from patient or legal representative.
* Subject of both genders (male and female not pregnant and not breastfeeding) aged over 49;
* Laboratory confirmation of 2019-nCoV infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source;
* Symptomatic subject with symptoms for up to 72 hours who does not require hospitalization, with signs and symptoms of acute respiratory viral infection characterized by a feverish sensation or fever, which may or may not be present at the time of the examination (which may be reported to the health professional), accompanied by cough or sore throat or runny nose or difficulty breathing and:

  i) Oxygen saturation ≥ 90%; ii) Risk classification for COVID-19 between low (A) or medium (B) (scores 1 to 19), according to the Brazilian Ministry of Health.

Exclusion Criteria:

* Participating in another RCT in the past 12 months;
* Presence of comorbidities, which have a contraindication to the use of the study product, not being restricted to:

  * HIV or HTLV virus infection;
  * Chronic hepatitis C (HCV) treated with direct antiviral drugs;
  * Liver failure;
  * Severe renal failure, including dialysis;
* Present hypersensitivity to the study product (nitazoxanide), as well as to related compounds;
* Concomitant administration of drugs that may interact with the product under study (nitazoxanide);
* Participants who underwent treatment with other antiviral drugs;
* Subject in antineoplastic treatment with chemotherapy or radiation therapy;
* Subject with severe autoimmune diseases in immunosuppression;
* Transplanted participants;
* Pregnant or lactating women;
* Any other clinical condition that is deemed by the Investigator to be an imminent risk to the health and life of the subject.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in signs and symptoms scale | 21 days
  Symptoms will be assessed using a 5 point scale (1- excellent, 2- good, 3- fair, 4 - poor 5 - very poor).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 21 days
  Number of participants with treatment-related adverse events
The proportion of subjects hospitalized after start of treatment and before the end of the study | 21 days
  Change in clinical condition - WHO Ordinal Scale for Clinical Improvement that measures illness severity over time (0=uninfected; ambulatory, no limitation of activities=1; ambulatory, limitation of activities=2, hospitalized no oxygen therapy=3; hospitalized oxygen by mask or nasal prongs=4; hospitalized non invasive ventilation or high-flow oxygen=5; hospitalized intubation or mechanical ventilation=6; hospitalized ventilation + additional organ support=7; death=8)
The proportion of subjects that need mechanical ventilation after start of treatment and before the end of the study | 21 days
  Change in clinical condition - WHO Ordinal Scale for Clinical Improvement that measures illness severity over time (0=uninfected; ambulatory, no limitation of activities=1; ambulatory, limitation of activities=2, hospitalized no oxygen therapy=3; hospitalized oxygen by mask or nasal prongs=4; hospitalized non invasive ventilation or high-flow oxygen=5; hospitalized intubation or mechanical ventilation=6; hospitalized ventilation + additional organ support=7; death=8)
Duration of symptoms | 21 days
  Time required (days) to full symptom recovery
Rate of mortality within 21-days | 21 days
  Evaluation of change in acute respiratory syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Edimilson Migowski, MD, Principal Investigator — NEPS SEMUS Mesquita

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.